CLINICAL TRIAL: NCT06110624
Title: The MuSt-PC: A Multidimensional Strategy to Improve Quality of Life of Patients With Multiple Symptoms and Palliative Care Needs - Feasibility Study
Brief Title: The MuSt-PC: a Feasibility Study on Intent to Use a Tool With Regard to Symptom Management
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 11265
Record Dates: First submitted 2023-10-07; First posted 2023-10-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Palliative Medicine
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arm 1: A targeted sample of healthcare providers (HCPs) who are not specialized in palliative care (GHCPs) constitutes the study population.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A survey study will be conducted to evaluate if GHCPs have the Intention to Use (IU) MuSt-PC in daily practice.

SUMMARY:
A study on the intent to use a tool (MuSt-PC) to manage symptoms of patients in a palliative care trajectory.

DETAILED DESCRIPTION:
A survey study will be conducted to evaluate if GHCPs have the Intention to Use (IU) MuSt- PC in daily practice. GHCPs are recruited via the connections of the seven Centers of Expertise in Palliative Care. To invite them to participate in the study, the GHCPs are approached directly via e-mail or telephone. Participating GHCPs will be educated on how to use MuSt-PC (educational materials and instruction webinar). GHCPs will be asked to use the CDSS for five individual patients. Every time after using MuSt-PC they will be asked to answer additional questions about their experience with using MuSt-PC in that specific instance. After using MuSt-PC for five patients, they are requested to fill out a comprehensive questionnaire about their overall experiences with using the CDSS.

ELIGIBILITY:
Inclusion Criteria:

Residents (in Dutch: Arts In Opleiding tot Specialist (AIOS) or Arts Niet In Opleiding tot Specialist (ANIOS)), medical specialists and nurse practitioners working in the following disciplines are invited to participate:

* General practice
* Nursing home
* Hospital:

  * Clinical geriatrics
  * Medical oncology
  * Radiation oncology
  * Pulmonology
  * Cardiology

Exclusion Criteria:

HCPs who were formally trained in palliative care ("kaderopleiding palliatieve zorg", "Masteropleiding Palliative Medicine for Health Care Professionals at Cardiff University" or "post-HBO opleiding palliatieve zorg") and/or who have been or are currently a consultant of a palliative care consultation team are considered specialists in palliative care, are excluded from participation.

GHCPs (e.g. nurses) who cannot independently decide about CDSS recommendation adherence, including drug interventions, are excluded from participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A targeted sample of healthcare providers (HCPs) who are not specialized in palliative care (GHCPs) constitutes the study population.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Questions evaluating Intention to Use (IU) | after 5 times use of the MuSt-PC tool within 3 months
  Questions evaluating Intention to Use (IU) (7-point Likert scales)

SECONDARY OUTCOMES:
Questions evaluating other modified TAM domains | after 5 times use of the MuSt-PC tool within 3 months
  Questions evaluating other modified TAM domains: Perceived Usefulness, Perceived Ease-of-Use, Attitude, Compatibility, Subjective norm, Facilitators, Habit (7-point Likert Scales).
Perceived benefits and disadvantages of using MuSt-PC | after 5 times use within 3 months
  Perceived benefits and disadvantages of using MuSt-PC (open-ended questions).
Suggestions to improve the MuSt-PC CDSS | after 5 times of the MuSt-PC tool within 3 months
  Suggestions to improve the MuSt-PC CDSS (open-ended question).
An overview of the content of questions of participating GHCPs regarding MuSt-PC use. | after 5 times use within 3 months
  An overview of the content of questions of participating GHCPs regarding MuSt-PC use. Questions will be analyzed qualitatively; coding will be done independently by two researchers. In case of disagreement, consensus will be achieved through discussion. Coding will result in categorization of question subject. Categorizations are ranked from most prevalent to least prevalent question subject (proportion of respondents).
Most useful elements of MuSt-PC will be evaluated with a multiple-choice question. | after 5 times use within 3 months
  Most useful elements of MuSt-PC will be evaluated with a multiple-choice question. (multiple answers allowed) Frequency and percentage of total respondents who chose the multiple choice answer possibilities will be evaluated
Mean scores of HCPs adherence to CDSS recommendations | after 5 times use of the MuSt-PC tool within 3 months
  Mean scores (5-point Likert scale) of HCPs adherence to CDSS recommendations (each time using MuSt-PC)

OTHER OUTCOMES:
A focus group meeting will be conducted if ≥20% of all participating GHCPs have insufficient intention to use MuSt-PC and/or perceive MuSt-PC insufficiently useful and/or perceive MuSt-PC insufficiently easy to use | after 5 times use of the MuSt-PC tool within 3 months
  A focus group meeting will be conducted if ≥20% of all participating GHCPs have insufficient intention to use MuSt-PC and/or perceive MuSt-PC insufficiently useful and/or perceive MuSt-PC insufficiently easy to use:
  1. Insufficient IU is defined as a sum score of ≤12 for the 3 questions that measure Intention to Use by the modified TAM questionnaire (maximum sum score 21)
  2. Insufficient PU is defined as a sum score of ≤24 for the 6 questions that measure PU by the modified TAM questionnaire (maximum sum score 42)
  3. insufficient PEU is defined as a sum score of ≤24 for the 6 items that measure PEU by the modified TAM questionnaire (maximum sum score 42). (see Appendix G) Six to twelve GHCPs with a sum score of ≤12 (IU) and/or ≤24 (PU and/or PEU) will be invited to participate.

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - LUMC, Leiden